CLINICAL TRIAL: NCT00798369
Title: An Adaptive Dose-ranging, Multi-center, Single-blind, Double-dummy, Active-controlled Trial to Determine the Target Dose of Canakinumab (ACZ885) in the Treatment of Acute Flares in Gout Patients Who Are Refractory or Contraindicated to NSAIDs and/or Colchicine
Brief Title: Targeted Dose Finding of Canakinumab (ACZ885) for Management of Acute Flare in Refractory or Contraindicated Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885H2255; EudraCT 2008-004666-61
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Acute Gout
Keywords: Acute flares; Gout; Anti-interleukin-1β monoclonal antibody; Colchicine; Triamcinolone acetonide
MeSH Terms: conditions — Gout | interventions — canakinumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Canakinumab 10 mg (Experimental): Canakinumab 10 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Canakinumab
- Canakinumab 25 mg (Experimental): Canakinumab 25 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Canakinumab
- Canakinumab 50 mg (Experimental): Canakinumab 50 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Canakinumab
- Canakinumab 90 mg (Experimental): Canakinumab 90 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Canakinumab
- Canakinumab 150 mg (Experimental): Canakinumab 150 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Canakinumab
- Triamcinolone acetonide 40 mg (Active Comparator): Triamcinolone acetonide 40 mg intramuscularly (i.m) once. The i.m. injection was recommended to be administered deeply into the gluteal muscle. Randomized patients received triamcinolone acetonide 40 mg i.m. once and placebo matching canakinumab s.c. once, on Day 1.
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Canakinumab — Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
  Arms: Canakinumab 10 mg
Drug: Canakinumab — Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1.
  Arms: Canakinumab 25 mg
Drug: Canakinumab — Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1.
  Arms: Canakinumab 50 mg
Drug: Canakinumab — Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1.
  Arms: Canakinumab 90 mg
Drug: Canakinumab — Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1.
  Arms: Canakinumab 150 mg
Drug: Triamcinolone acetonide — Randomized patients received triamcinolone acetonide 40 mg i.m. once and placebo matching canakinumab s.c. once, on Day 1.
  Arms: Triamcinolone acetonide 40 mg

SUMMARY:
This 8-week study is designed to determine the target dose of canakinumab (ACZ885) for the management of acute flare in gout patients who are contraindicated to Non-Steroidal anti-inflammatory drugs and/or colchicine. The efficacy of ACZ885 will be compared to the corticosteroid triamcinolone acetonide.

ELIGIBILITY:
Inclusion Criteria:

* History of at least 1 gout flare prior to the Screening Visit
* Meeting the American College of Rheumatology (ACR) 1977 preliminary criteria for the classification of acute arthritis of primary gout.
* Presence of acute gout flare for no longer than 5 days.
* Baseline pain intensity > or = to 50 mm on the 0-100 mm VAS.
* Contraindicated for, intolerant or unresponsive to NSAIDs, colchicine or both.

Exclusion Criteria:

* Rheumatoid arthritis, evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis.
* Presence of severe renal function impairment
* Contraindication to intramuscular injection
* Known presence or suspicion of active or recurrent bacterial, fungal or viral infection at the time of enrollment
* Evidence of active pulmonary disease
* Live vaccinations within 3 months prior to the start of the study
* Use of forbidden therapy

Other protocol-defined inclusion/exclusion criteria applied

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (27):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Associated Pharmaceutical Research, Buena Park, California
  - Northern California Institute for Bone Health, Oakland, California
  - San Diego Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Tampa Medical Group, P.A., Tampa, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Harbin Clinic, Rome, Georgia
  - Intermountain Orthopedics, Boise, Idaho
  - Northwest Clinical Trials, Boise, Idaho
  - The Arthritis Center, Springfield, Illinois
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Montana Medical Research, Missoula, Montana
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Regional Clinical Research Rheumatology Assoc., Binghamton, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Community Research Partners, Inc., Varnville, South Carolina
  - Comprehensive Rheumatology, Hendersonville, Tennessee
  - MultiSpecialty Clinical Research, Johnson City, Tennessee
  - Integrity Clinical Research, LLC, Milan, Tennessee
  - Southwest Rheumatology, Mesquite, Texas
  - Health Research of Hampton Roads, Newport News, Virginia
- Novartis Investigative site, Rosario, Argentina
- Novartis Investigative site, Gozée, Belgium
- Canada (3):
  - Novartis Investigative site, Moncton
  - Novartis Investigative site, Mount Pearl
  - Novartis Investigative site, St. John's
- Novartis Investigative site, Paris, France
- Germany (16):
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Bautzen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dachau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Georgensgmünd
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Messkirch
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, Schwabach
  - Novartis Investigative Site, Zerbst
- Poland (3):
  - Novartis Investigative site, Poznan
  - Novartis Investigative site, Szczecin
  - Novartis Investigative site, Wroclaw
- Russia (6):
  - Novartis Investigative site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative site, Tyumen
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative site, Yekaterinburg
- Switzerland (4):
  - Novartis Investigative site, Baden
  - Novartis Investigative site, Basel
  - Novartis Investigative site, Bern
  - Novartis Investigative site, Lausanne
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Manisa
  - Novartis Investigative site, Sihhiye/Ankara
- United Kingdom (4):
  - Novartis Investigative Site, Antrim
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, Wellingborough

REFERENCES:
- [Derived] Chakraborty A, Van LM, Skerjanec A, Floch D, Klein UR, Krammer G, Sunkara G, Howard D. Pharmacokinetic and pharmacodynamic properties of canakinumab in patients with gouty arthritis. J Clin Pharmacol. 2013 Dec;53(12):1240-51. doi: 10.1002/jcph.162. Epub 2013 Sep 30. PMID 24122883
- [Derived] Schlesinger N, De Meulemeester M, Pikhlak A, Yucel AE, Richard D, Murphy V, Arulmani U, Sallstig P, So A. Canakinumab relieves symptoms of acute flares and improves health-related quality of life in patients with difficult-to-treat Gouty Arthritis by suppressing inflammation: results of a randomized, dose-ranging study. Arthritis Res Ther. 2011 Mar 25;13(2):R53. doi: 10.1186/ar3297. PMID 21439048
- [Derived] So A, De Meulemeester M, Pikhlak A, Yucel AE, Richard D, Murphy V, Arulmani U, Sallstig P, Schlesinger N. Canakinumab for the treatment of acute flares in difficult-to-treat gouty arthritis: Results of a multicenter, phase II, dose-ranging study. Arthritis Rheum. 2010 Oct;62(10):3064-76. doi: 10.1002/art.27600. PMID 20533546

RESULTS

PARTICIPANT FLOW:
Groups:
- Canakinumab 10 mg: Canakinumab 10 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once,on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
- Canakinumab 25 mg: Canakinumab 25 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once,on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
- Canakinumab 50 mg: Canakinumab 50 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once,on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
- Canakinumab 90 mg: Canakinumab 90 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once,on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
- Canakinumab 150 mg: Canakinumab 150 mg subcutaneous (s.c) once. The s.c. injection could be administered into the arm or thigh. Randomized patients received one s.c. injection of canakinumab and placebo matching triamcinolone acetonide (0.9% sodium chloride) intramuscularly (i.m.) once,on Day 1. The i.m. injection was recommended to be administered deeply into the gluteal muscle.
- Triamcinolone Acetonide 40 mg: Triamcinolone acetonide 40 mg intramuscularly (i.m) once. The i.m. injection was recommended to be administered deeply into the gluteal muscle. Randomized patients received triamcinolone acetonide 40 mg i.m. once or canakinumab matching placebo once, on Day 1.
Period: Overall Study
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 28 | 29 | 29 | 29 | 28 | 57
Completed | 27 | 28 | 27 | 28 | 27 | 54
Not Completed | 1 | 1 | 2 | 1 | 1 | 3
Not completed — Subject withdrew consent | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 1 | 0
Not completed — Adminstrative problems | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg | Total
Number analyzed (Participants) | 28 | 29 | 29 | 29 | 28 | 57 | 200
Age, Customized [Number; unit: participants]
  ≥18 years - 40 years | 6 | 4 | 3 | 5 | 8 | 7 | 33
  ≥ 41 - 64 years | 21 | 21 | 19 | 20 | 15 | 39 | 135
  ≥ 65 - 74 years | 0 | 3 | 6 | 2 | 3 | 10 | 24
  ≥ 75 years | 1 | 1 | 1 | 2 | 2 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 5 | 0 | 2 | 14
  Male | 26 | 26 | 27 | 24 | 28 | 55 | 186

OUTCOME MEASURES:

1. Secondary Outcome: The Change in Pain Intensity in the Target Joint Following Canakinumab Administration Compared to Triamcinolone Acetonide
Description: The change in pain intensity from baseline to 72 hours and 7 days post dose as measured on a 0-100 mm Visual Analog Scale(VAS): 0= no pain and 100= severe pain. Analysis of Covariance (ANCOVA) with treatment group, VAS at baseline and Body mass Index (BMI) at baseline as covariates. Change from baseline = (post-baseline measurement - baseline).
Time Frame: Baseline,at 72 hrs post-dose and 7 days post-dose
Population: Full Analysis Set consisting of all participants with data for baseline and the given time point for each arm/group. Assessments up to Day 8, with 1 missing pain intensity value had it imputed. LOCF method was applied to impute post-dose measurements. Missing baseline values were replaced by the median baseline assessment
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 28 | 29 | 28 | 29 | 27 | 56
Units on a scale
  72 hrs post-dose (n= 28, 28, 26, 28, 27, 53) | -48.6 (4.36) | -46.6 (4.39) | -48.6 (4.56) | -52.7 (4.35) | -62.5 (4.58) | -43.3 (3.16)
  7 days post-dose (n= 26, 28, 27, 27, 26, 51) | -57.6 (4.06) | -53.9 (3.93) | -63.4 (4.00) | -61.2 (3.96) | -66.4 (4.19) | -56.0 (2.88)

2. Secondary Outcome: Percentage of Participants With an Excellent or Good Response With Regards to the Patient's Global Assessment of Response to Treatment
Description: Participants scored their global assessment of response to treatment using a 5-point Likert scale: Excellent, Good, Acceptable, Slight and Poor.
Time Frame: at 72 hours post-baseline
Population: The Full Analysis Set (FAS) consisted of all participants as randomized that had at least one post-baseline assessment of the primary efficacy variable. Following the intent-to-treat principle, participants were analyzed according to the treatment they were assigned to at randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 28 | 29 | 28 | 29 | 27 | 56
Percentage of Participants | 64 | 62 | 71 | 66 | 89 | 54

3. Secondary Outcome: The Time to 50% Reduction of Baseline Pain Intensity in the Target Joint
Description: The median time in days to at least 50% reduction in Pain intensity from baseline as measured by Visual Analog Scale (VAS) for each treatment group. Participants scored their pain intensity in the target joint on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100).
Time Frame: Baseline, within 7 days after randomization
Population: The Full Analysis Set (FAS) consisted of all participants as randomized that had at least one post baseline assessment of the primary efficacy variable. Following the intent-to-treat principle, participants were analyzed according to the treatment they were assigned to at randomization.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 28 | 29 | 28 | 29 | 27 | 56
Days | 2.9 [1.0 to 4.0] | 2.9 [2.0 to 3.0] | 1.0 [1.0 to 2.9] | 1.0 [1.0 to 2.0] | 1.0 [0.5 to 2.0] | 2.0 [1.0 to 3.6]

4. Secondary Outcome: High Sensitivity C-reactive Protein (hsCRP) at 72 Hours, 7days, 4 Weeks and 8 Weeks Post Dose for Each Treatment Group
Description: High sensitivity C-reactive protein (hsCRP) was determined in serum at all visits (Visits 1-5) in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.
  ANCOVA with treatment group, protein level at baseline and BMI at baseline as covariates.
Time Frame: at 72 hours and 7 days, 4 and 8 weeks post-dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 28 | 29 | 28 | 29 | 27 | 56
mg/L
  72 hrs post-dose (n= 27, 28, 26, 28, 25, 53) | 16.7 (3.41) | 7.9 (3.34) | 11.7 (3.49) | 13.4 (3.34) | 9.2 (3.53) | 13.4 (2.43)
  7 days post-dose (n= 28, 29, 28, 28, 27, 55) | 8.0 (3.30) | 2.5 (3.23) | 4.3 (3.31) | 6.3 (3.29) | 3.7 (3.36) | 13.7 (2.35)
  4 week post-dose (n= 27, 28, 27, 28, 27, 55) | 3.0 (3.13) | 2.9 (3.08) | 2.9 (3.14) | 4.8 (3.08) | 4.8 (3.13) | 9.2 (2.20)
  8 weeks post-dose (n= 26, 28, 27, 28, 27, 54) | 3.8 (1.79) | 2.0 (1.72) | 2.6 (1.75) | 5.2 (1.72) | 2.9 (1.75) | 8.6 (1.24)

5. Secondary Outcome: Serum Amyloid Protein (SAA) Levels at 72 Hours, 7days, 4 Weeks and 8 Weeks Post Dose for Each Treatment Group
Description: Serum amyloid A (SAA) were determined in serum at all visits (Visits 1-5) in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.
  ANCOVA with treatment group, protein level at baseline and BMI at baseline as covariates.
Time Frame: at 72 hours and 7 days, 4 and 8 weeks post-dose
Population: The Full Analysis Set (FAS) consisted of all patients as randomized that had at least one post-baseline assessment of the primary efficacy variable. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 28 | 29 | 28 | 29 | 27 | 56
mg/L
  72 hrs post-dose (n= 26, 28, 28, 28, 27, 50) | 50.1 (20.05) | 27.6 (19.32) | 70.7 (19.37) | 29.4 (19.28) | 26.9 (19.69) | 52.5 (14.48)
  7 days post-dose (n= 28, 28, 28, 28, 26, 49) | 10.6 (10.92) | 5.4 (10.91) | 11.9 (10.94) | 10.5 (10.89) | 10.3 (11.33) | 39.4 (8.26)
  4 week post-dose (n= 27, 28, 27, 28, 27, 50) | 4.4 (3.53) | 4.2 (3.46) | 4.9 (3.53) | 14.3 (3.45) | 6.2 (3.53) | 12.9 (2.59)
  8 weeks post-dose (n= 26, 26, 26, 27, 27, 48) | 5.5 (3.64) | 4.6 (3.64) | 5.7 (3.64) | 8.2 (3.56) | 4.1 (3.57) | 18.0 (2.68)

6. Primary Outcome: The Dose of Canakinumab for Treatment of Acute Flares in Gout Patients That Leads to the Same Efficacy as Triamcinolone Acetonide With Respect to Pain Intensity on a 0-100 mm Visual Analog Scale (VAS)
Description: Mean target dose at 24, 48 and 72 hours. Four models: Emax, Logistic, Linear in log-dose, Linear were selected to describe the potential dose-response curve and hence estimate the target dose of canakinumab using baseline Visual Analog Scale (VAS) and Body Mass Index (BMI) as covariates. Target dose was defined as the dose for which the efficacy is equivalent to the efficacy of triamcinolone acetonide 40 mg and was identified by assessing the dose response relationship with regards to the pain intensity in the target joint measured on a 0- 100 mm VAS (0= no pain and 100= unbearable pain).
Time Frame: at 24,48 and 72 hours post-baseline
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: mg
Groups:
- Linear Model: The linear model was the best-fitting model out of the 4 selected models (Emax, Logistic, Linear in Log-dose, Linear)with lowest Akaike Information Criterion (AIC).
Arm/Group | Linear Model
Number analyzed (Participants) | 197
mg
  Target dose at 24 hrs post-baseline | 37 [5.94 to 103.37]
  Target dose at 48 hrs post-baseline | 23 [2.87 to 96.31]
  Target dose at 72 hrs post-baseline | NA [NA to NA] — A target dose for canakinumab to be comparable to triamcinolone acetonide 40 mg could not be estimated at 72 hours as it lies below the range of all doses of canakinumab tested in this trial

7. Secondary Outcome: Amount of Rescue Medication Taken for Each Treatment Group
Description: Participants who had difficulty in tolerating their pain after the 6-hour post-dose pain assessments and during the first 7 study days were allowed to take a maximum of 30 mg prednisolone (or equivalent dose of prednisone [30 mg]) orally once a day for a maximum of 5 days. In addition, participants could use 500 mg acetaminophen (paracetamol) and/or 30 mg codeine as needed during the first 7 study days. A maximum of 1 g/dose or 3 g/day of acetaminophen and 30 mg/dose or 180 mg/day of codeine was allowed during the first 7 days of the study.
Time Frame: 7 days after study drug administration
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 28 | 29 | 28 | 29 | 27 | 56
mg
  Acetaminophen | 1414.3 (2628.58) | 1656.9 (4437.26) | 2178.6 (2925.67) | 1646.6 (3161.20) | 607.4 (2250.12) | 1614.3 (2958.51)
  Codeine | 42.9 (138.19) | 78.6 (164.20) | 49.3 (139.57) | 27.9 (87.07) | 4.4 (23.09) | 52.0 (158.28)
  Prednisolone/Prednisone | 13.4 (36.82) | 23.8 (44.03) | 24.1 (59.36) | 13.1 (35.37) | 6.2 (24.54) | 13.3 (26.13)

ADVERSE EVENTS:
Time Frame: End of study (8 weeks)
Arm/Group | Canakinumab 10 mg | Canakinumab 25 mg | Canakinumab 50 mg | Canakinumab 90 mg | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Serious Adverse Events (participants affected / at risk) | 0/28 | 2/29 | 2/29 | 0/29 | 0/28 | 1/57
Other Adverse Events (participants affected / at risk) | 2/28 | 7/29 | 5/29 | 8/29 | 5/28 | 8/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 10 mg (N=28) | Canakinumab 25 mg (N=29) | Canakinumab 50 mg (N=29) | Canakinumab 90 mg (N=29) | Canakinumab 150 mg (N=28) | Triamcinolone Acetonide 40 mg (N=57)
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 10 mg (N=28) | Canakinumab 25 mg (N=29) | Canakinumab 50 mg (N=29) | Canakinumab 90 mg (N=29) | Canakinumab 150 mg (N=28) | Triamcinolone Acetonide 40 mg (N=57)
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 3
Headache (Nervous system disorders) | 1 | 3 | 1 | 2 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.